CLINICAL TRIAL: NCT01167608
Title: Barriers to Mental Healthcare Utilization in Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Roseanne D Dobkin, PhD, Associate Professor, Rutgers, The State University of New Jersey
Other Study IDs: 0220100120; 1K23NS052155-01A2 (NIH)
Record Dates: First submitted 2010-07-20; First posted 2010-07-22 (Estimated); Results first posted 2014-07-04 (Estimated); Last update posted 2019-07-16 (Actual); Status verified 2019-06

CONDITIONS: Parkinson's Disease; Depression; Anxiety
Keywords: Parkinson's disease; Depression; Anxiety; Treatment
MeSH Terms: conditions — Parkinson Disease; Depression; Anxiety Disorders

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- People with Parkinson's disease: Individuals diagnosed with Parkinson's disease
  Interventions: Other: No Intervention. This is a cross-sectional survey study.

INTERVENTIONS:
Other: No Intervention. This is a cross-sectional survey study. — No intervention.

SUMMARY:
Parkinson's disease (PD) is the second most common neurodegenerative disorder in the elderly. In most people, the illness is complicated by co-occurring psychiatric problems such as depression and anxiety. These non-motor concerns negatively affect the course and management of the disease, often leading to poor outcomes for both patients and their families. Despite these deleterious consequences, psychiatric symptoms in PD are both underreported by patients as well as under-recognized and under-treated by health care providers.

The primary purpose of this study is to identify and describe barriers to mental healthcare utilization for people with Parkinson's disease. Secondary objectives include the assessment of attitudes and preferences regarding the need for mental health services in the PD community and the acceptability of telehealth interventions as a method for improving access and quality of care. In order to accomplish these aims, participants will be asked to fill out an anonymous survey which will take about 15-30 minutes to complete. To best accommodate PD patients with varying levels of disability, participants will have the option to complete the survey online, on paper, or over the phone. The information obtained from this study will be used to support future treatment development efforts (i.e., phone and internet based interventions, community based trainings with local providers) intended to improve access and quality of mental health care for people with PD. To the best of the investigators knowledge, this is the first study to systematically examine barriers to mental healthcare utilization in PD in a national sample.

DETAILED DESCRIPTION:
The survey may be completed online at https://www.surveymonkey.com/s/improvecare4pd. Potential participants may also call Dr. Dobkin at 732-235-4051 to complete the survey over the phone or to request a paper copy to mailed out.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Parkinson's disease
* At least 18 years of age

Exclusion Criteria:

* Less than 18 years of age

We are looking for responses from those who have, as well as those who have not, had mental health treatment in the past.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People with Parkinson's disease.
Sampling Method: Probability Sample
Enrollment: 883 (Actual)
Dates: Start 2010-06; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roseanne D Dobkin, PhD, Principal Investigator — Rutgers, The State University of New Jersey
Locations (1):
- Rutgers-Robert Wood Johnson Medical School, Piscataway, New Jersey, United States

REFERENCES:
- [Result] Dobkin RD, Rubino JT, Friedman J, Allen LA, Gara MA, Menza M. Barriers to mental health care utilization in Parkinson's disease. J Geriatr Psychiatry Neurol. 2013 Jun;26(2):105-16. doi: 10.1177/0891988713481269. Epub 2013 Apr 15. PMID 23589410

RESULTS

PARTICIPANT FLOW:
Recruitment Details: People with Parkinson's disease throughout the United States (US) were recruited from several sources (i.e., support groups affiliated with the American Parkinson's disease Association; internet sites such as the Michael J. Fox Foundation Fox Trial Finder Wedsite). Recruitment took place between June of 2010 and February of 2012.
Groups:
- People With Parkinson's Disease: No Intervention. This is a cross-sectional survey study. : No intervention.
Period: Overall Study
Arm/Group | People With Parkinson's Disease
Started | 883
Completed | 769
Not Completed | 114

BASELINE CHARACTERISTICS:
Arm/Group | People With Parkinson's Disease
Number analyzed (Participants) | 883
Age, Customized [Number; unit: participants]
  <=18 years | 0
  Between 18 and 65 years | 408
  >=65 years | 347
  Not Available | 128
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.83 (10.45)
Sex/Gender, Customized [Number; unit: participants]
  Female | 375
  Male | 380
  Not Available | 128
Region of Enrollment [Number; unit: participants]
  United States | 883

OUTCOME MEASURES:

1. Primary Outcome: Most Commonly Reported Past Barrier to Mental Health Services: "Anyone in my Situation Would be Struggling"
Description: The purpose of this study was to assess the 3 most commonly reported past and future barriers to mental health services. This outcome represents the most common past barrier to mental health services reported by survey respondents. The outcome reported is the percentage of all respondents surveyed who endorsed this particular past barrier. This barrier can best be described as low mental health literacy.
Time Frame: Baseline
Population: This is an anonymous, cross-sectional survey study. Not all participants responded to every item, so sample size varies between outcome measures.
Measure: Number; unit: percentage of total respondents
Arm/Group | People With Parkinson's Disease
Number analyzed (Participants) | 103
percentage of total respondents | 74.8

2. Primary Outcome: 2nd Most Commonly Reported Past Barrier to Mental Health Services: "Doctors Are Not Sensitive Enough to PD-related Issues"
Description: The purpose of this study was to assess the 3 most commonly reported past and future barriers to mental health services. This outcome represents the 2nd most common past barrier to mental health services reported by survey respondents. The outcome reported is the percentage of all respondents surveyed who endorsed this particular past barrier. This barrier can best be described as limited knowledge of PD amongst treatment providers.
Time Frame: Baseline
Population: as for outcome 1
Measure: Number; unit: percentage of total respondents
Arm/Group | People With Parkinson's Disease
Number analyzed (Participants) | 104
percentage of total respondents | 54.8

3. Primary Outcome: 3rd Most Commonly Reported Past Barrier to Mental Health Services: "Out of Pocket Cost Was Too High"
Description: The purpose of this study was to assess the 3 most commonly reported past and future barriers to mental health services. This outcome represents the 3rd most common past barrier to mental health services reported by survey respondents. The outcome reported is the percentage of all respondents surveyed who endorsed this particular past barrier. This barrier can best be described as limited access.
Time Frame: Baseline
Population: as for outcome 1
Measure: Number; unit: percentage of total respondents
Arm/Group | People With Parkinson's Disease
Number analyzed (Participants) | 103
percentage of total respondents | 40.8

4. Primary Outcome: Most Commonly Reported Future Barrier to Mental Health Services: "Out of Pocket Cost Was Too High"
Description: The purpose of this study was to assess the 3 most commonly reported past and future barriers to mental health services. This outcome represents the most common future barrier to mental health service reported by respondents to the survey described in the Methods section. Outcome is reported as the percentage of all respondents surveyed who endorsed this particular future barrier. This barrier can best be described as limited access.
Time Frame: Baseline
Population: as for outcome 1
Measure: Number; unit: percentage of total respondents
Arm/Group | People With Parkinson's Disease
Number analyzed (Participants) | 659
percentage of total respondents | 64.0

5. Primary Outcome: 2nd Most Commonly Reported Future Barrier to Mental Health Services: "Doctors Are Not Sensitive Enough to PD-related Issues"
Description: The purpose of this study was to assess the 3 most commonly reported past and future barriers to mental health services. This outcome represents the 2nd most commonly reported future barrier to mental health services reported by those who responded to the survey described in the Methods section. Outcome is reported as the percentage of all respondents surveyed who endorsed this particular future barrier. This barrier can best be described as limited knowledge of PD amongst treatment providers.
Time Frame: Baseline
Population: as for outcome 1
Measure: Number; unit: percentage of total respondents
Arm/Group | People With Parkinson's Disease
Number analyzed (Participants) | 658
percentage of total respondents | 58.7

6. Primary Outcome: 3rd Most Commonly Reported Future Barrier to Mental Health Services: "Services Are Not Available in my Community"
Description: The purpose of this study was to assess the 3 most commonly reported past and future barriers to mental health services. This outcome represents the 3rd most common future barrier to mental health service reported by respondents to the survey described in the Methods section. Outcome is reported as the percentage of all respondents surveyed who endorsed this particular future barrier. This barrier can best be described as limited access.
Time Frame: Baseline
Population: as for outcome 1
Measure: Number; unit: percentage of total respondents
Arm/Group | People With Parkinson's Disease
Number analyzed (Participants) | 661
percentage of total respondents | 52.0

ADVERSE EVENTS:
Arm/Group | People With Parkinson's Disease
Serious Adverse Events (participants affected / at risk) | 0/769
Other Adverse Events (participants affected / at risk) | 0/769

LIMITATIONS AND CAVEATS:
Self-report biases (social desirability or recall); idiopathic PD could not be confirmed given the anonymous nature of study participation; results may not generalize to all people with PD; participants were self-selected (non-random sample)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes